CLINICAL TRIAL: NCT06245109
Title: Brain-Based and Clinical Phenotyping of Pain Pharmacotherapy in Knee Osteoarthritis
Acronym: PREDICT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Thomas J. Schnitzer, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: STU00219434
Record Dates: First submitted 2024-01-29; First posted 2024-02-07 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
Keywords: knee oa; knee osteoarthritis; osteoarthritis; knee pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Duloxetine Hydrochloride; Celecoxib

STUDY DESIGN:
Intervention Model Description: Synopsis of study design:
  The goal of this study is to identify predictors of treatment response, using quantitative sensory testing (QST), neuroimaging, and patient-reported outcome measures (PROs).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Duloxetine (Active Comparator): Duloxetine 60mg tablet, daily (with an initial and final 7-day titration at 30 mg, daily)
  Interventions: Drug: Duloxetine
- Celecoxib (Active Comparator): Celecoxib 200 mg tablet, daily
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator): Matching placebo tablet, daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — 60 mg, oral
  Other Names: Cymbalta
  Arms: Duloxetine
Drug: Celecoxib — 200 mg, oral
  Other Names: Celebrex
  Arms: Celecoxib
Drug: Placebo — Matching placebo, oral
  Arms: Placebo

SUMMARY:
This is a clinical trial of people who have pain due to knee osteoarthritis at Northwestern University Feinberg School of Medicine. The study will last for about 20 weeks. 180 qualified participants will be randomly assigned in a 1:1:1 ratio (60 participants per group) to one of three treatment groups: duloxetine, celecoxib, or placebo. Participants will have an Xray, knee MRI, brain MRI, blood draws, pain sensitivity testing, and asked to fill out questionnaires. The purpose of this study is to try to predict which participants will respond to the treatment.

DETAILED DESCRIPTION:
This longitudinal study will screen and enroll 180 participants diagnosed with knee osteoarthritis at Northwestern University Feinberg School of Medicine. The study will last for about 20 weeks' duration with a repeat-treatment design. An equal number of participants (60 per group) will be randomly assigned in a 1:1:1 ratio, stratified by sex and current opioid use, to one of three treatment groups after they qualify to enter the study. The treatment groups will celecoxib (200 mg qd), duloxetine (60 mg qd, with an initial and final 7-day titration at 30 mg qd), or matching placebo (one capsule qd). This aim of this study is to identify specific biomarkers in individual people with knee osteoarthritis pain that will allow definition of responder phenotypes distinct for different therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age greater than 40 years, with no racial/ethnic restrictions;
2. Meet American College of Radiology (ACR) criteria for knee osteoarthritis (OA) based on radiographic evidence;
3. Knee pain most days of the week for the past month at screening;
4. Must have average pain score for the week prior to baseline of ≥ 4 (on a 0 to 10 NRS)
5. Must complete pain ratings on at least 4 out of 7 days prior to baseline
6. Must be able to read and speak English and be willing to read and understand instructions as well as questionnaires;
7. Must be in generally stable health;
8. Must be able to return for all clinic visits;
9. Willing to remain stable on any concomitant therapies (TENs unit, ice, glucosamine chondroitin, cannabinoids, etc.)
10. Must sign an informed consent document after complete explanation of the study documenting that they understand the purpose of the study, procedures to be undertaken, possible benefits, potential risks, and are willing to participate.
11. Ambulatory with or without a cane, brace(s), or walking stick (use of walker or wheelchair will be exclusionary)

Exclusion Criteria:

1. Evidence of rheumatoid arthritis, ankylosing spondylitis, other inflammatory arthropathy;
2. Functional class IV congestive heart failure;
3. Significant other medical disease such as uncontrolled hypertension, untreated diabetes mellitus, coronary or peripheral vascular disease, chronic obstructive lung disease, liver disease (Liver Function Tests >3x Upper limit of normal) or malignancy;
4. Current use of illicit drugs or history (in last 12 months) of alcohol or drug abuse;
5. Current cannabinoid use for knee pain;
6. High dose opioid use, as defined as > 50mg morphine equivalent/day;
7. Any medical condition that in the investigator's judgment may prevent the individual from completing the study or put the individual at undue risk;
8. In the judgment of the investigator, unable or unwilling to follow protocol and instructions;
9. Intra-axial implants (e.g., spinal cord stimulators or pumps);
10. All exclusion criteria for Magnetic Resonance Imaging (MRI) safety: any metallic implants, brain or skull abnormalities, tattoos on large body parts, and claustrophobia;
11. Currently breastfeeding, pregnant, or planning to become pregnant during the study;
12. Chronic neurologic conditions, e.g., Parkinson's;
13. Renal insufficiency (creatinine >1.5 mg/dl)
14. Previous history of peptic ulcer or gastrointestinal bleeding
15. Current use of anticoagulants or platelet inhibitors other than aspirin (ASA) at ≤325 mg/day
16. Allergy to sulfonamide drugs, duloxetine, NSAIDs, or acetaminophen
17. Acute myocardial infarction or coronary artery bypass graft surgery, in the past 12 months
18. Recent injection into the index knee of hyaluronic acid or other substance in the last 6 months, or steroid in the last 90 days.
19. Severe lactose intolerance
20. Current use of selective serotonin reuptake inhibitors (SSRIs), serotonin and norepinephrine reuptake inhibitors (SNRIs), and/or tricyclic antidepressants (TCAs) at a therapeutic dose. Occasional use of these medications as a sleep aid will be allowed; however, participants will need to agree to remain on a stable dose of the medication while in the study.
21. Uncontrolled narrow-angle glaucoma

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Individuals with at least 30% Pain Response to treatment | Baseline to end of first treatment period (week 6) and second treatment period (week 16)
  At least 30% improvement from baseline in "weekly average daily pain" measured using a numeric rating scale (0-10) with 0 = no pain and 10 = worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Schnitzer, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States